CLINICAL TRIAL: NCT06227403
Title: Can A Youth Leadership and Mindfulness Program Support Well-being in Adolescence?
Brief Title: Leadership, Engagement, and Youth Action Program With Mindfulness (LEAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Massachusetts General Hospital (Other); University of Illinois at Chicago (Other); Utah State University (Other)
Responsible Party: Principal Investigator, Jennifer Greif Green, Professor, Wheelock College of Education & Human Development, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1UG3AT012530-01 (NIH)
Record Dates: First submitted 2024-01-05; First posted 2024-01-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Adolescent Behavior; Mental Health Wellness 1
Keywords: mindfulness; youth leadership; youth wellbeing
MeSH Terms: conditions — Adolescent Behavior | interventions — Leadership; Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leadership, Engagement, and youth Action Program with Mindfulness (Experimental): The Leadership, Engagement, and youth Action Program with Mindfulness intervention (LEAP) consists of 14 sessions focused on youth leadership and mindfulness.
  Interventions: Behavioral: Leadership, Engagement, and youth Action Program with Mindfulness
- EnvisionIT (Active Comparator): EnvisionIT is a college and career-readiness program designed for students in grades 6-12. The EnvisionIT program will be delivered over 14 sessions, and focus on skills and career/college readiness.
  Interventions: Behavioral: EnvisionIT

INTERVENTIONS:
Behavioral: Leadership, Engagement, and youth Action Program with Mindfulness — The Leadership, Engagement, and youth Action Program with Mindfulness intervention (LEAP) was designed and co-created with youth to improve youth well-being by enhancing leadership opportunities and by developing mindfulness in day-to-day life. LEAP seeks to foster these improvements in youth as a strategy to increase mental, emotional, and behavioral health. Youth voice is incorporated into the intervention, with facilitators leading the first 7 sessions, and youth leading the remainder.
  Arms: Leadership, Engagement, and youth Action Program with Mindfulness
Behavioral: EnvisionIT — Participants in this arm will receive 14 sessions of EnvisionIT training, focused on preparing students with essential skills including digital literacy through competency in information technology, financial literacy, English language arts skills, and college and career readiness. All sessions will be delivered by facilitators trained in EnvisionIT.
  Arms: EnvisionIT

SUMMARY:
The current study tests the feasibility and effectiveness of a youth intervention designed to provide meaningful leadership opportunities through the acquisition of leadership skills as well as mindfulness practice, LEAP: Leadership, Engagement, and youth Action Program with Mindfulness.

The goal of our proposal is to determine whether the Leadership, Engagement, and youth Action Program with Mindfulness (LEAP) curriculum, which was developed with youth, is a feasible and effective intervention for fostering leadership and well-being. We seek to understand whether LEAP can support well-being for youth as a strategy to increase youth mental, emotional, and behavioral (MEB) health.

DETAILED DESCRIPTION:
The LEAP study will determine whether a 14-session program designed to provide leadership and mindfulness skills to youth is an effective and feasible intervention. The curriculum consists of 14 two-hour sessions delivered after school. The comparison group will take part in EnvisionIT, a college and career readiness program designed for students in grades 6 through 12. EnvisionIT aims to prepare students with essential skills including digital literacy, and college and career readiness. The comparison group will also have 14 two-hour group sessions. Both LEAP and EnvisionIT will be delivered by trained facilitators. All participants in LEAP and EnvisionIT will be assessed at two time points assessing program outcomes; facilitators will also complete interviews post-intervention and provide feedback on data fidelity and acceptability following each session. This record reports on the UG3 pilot phase and will be amended for a UH3 phase.

ELIGIBILITY:
Inclusion Criteria:

• Adolescents ages 14-18 in grades 9-12 enrolled in collaborating sites, either in Massachusetts or Illinois.

Exclusion Criteria:

* Adolescents who are not available to commit to the intervention schedule.
* Adolescents who are not in grades 9-12.
* Parents/guardians with preferred language other than English or Spanish.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Mental Health Continuum - Short Form | Baseline, 2-3 months
  14-item, 6-point scale that measures emotional, social, and psychological wellbeing through frequency of experiencing each symptom of positive mental health. The scale range is 0-70, higher scores indicate better mental health.
Engagement, Perseverance, Optimism, Connectedness, and Happiness (EPOCH) measure of adolescent wellbeing | Baseline, 2-3 months
  20-item, 5-point scale measuring five positive characteristics that support higher levels of wellbeing: Engagement, Perseverance, Optimism, Connectedness, and Happiness. The scale range is 1-5, higher scores indicate better wellbeing.
Social Emotional Health Survey: Belief in Self-Domain | Baseline, 2-3 months
  9 item, 4-point measure of core psychological assets, measuring self-efficacy, self-awareness, and persistence. The scale range is 9-36, higher scores indicate better social emotional health.
Strengths and Difficulties Questionnaire | Baseline, 2-3 months
  25 item multiple choice questionnaire that measures internalizing and externalizing problems and prosocial behavior (emotional, conduct, hyperactivity-inattention, peer, prosocial). The scale range is 0-40, higher scores indicate worse difficulties.
Self-Rated Health | Baseline, 2-3 months
  12 item 5-point survey measuring general health, asking about overall health self-rating, ability to do daily activities, energy levels, and physical and emotional limitations. The scale range is 0-100, higher scores indicate better health.
Student Career Construction Inventory | Baseline, 2-3 months
  An 18 item, 4-point scale measuring ability to crystallize vocational self-concepts, explore information gathering about occupations, and preparing to implement that choice. The scale range is 1-5, higher scores indicate better career outcomes.
Vocational Skills Self-Efficacy | Baseline, 2-3 months
  A 37 item, 5-point scale that measures vocational competency. The scale range is 1-5, higher scores indicate better vocational skills self-efficacy.
Information and Communications Technology (ICT) Literacy Pretest-Posttest | Baseline, 2-3 months
  A 35 item multiple choice questionnaire that measures understanding of tools/mechanics of the internet, research processes, and application to career research. The scale range is 0-29, higher scores indicate better ICT literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer G Green, PhD, Principal Investigator — Boston University; Mario Cruz-Gonzalez, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - University of Illinois Chicago, Chicago, Illinois
  - METCO, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Data for the study UG3 Phase are for pilot and feasibility purposes and will not be shared with other researchers.